CLINICAL TRIAL: NCT01669460
Title: A Phase II, Open Label Study of Red Bull™ Sugar-Free Drink for Reduction of Fatigue in Prostate Cancer Patients Receiving LHRH Agonist Therapy
Brief Title: Study of Red Bull™ Sugar-Free Drink for Reduction of Fatigue in Prostate Cancer Patients Receiving LHRH Agonist Therapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 12-5041-C
Record Dates: First submitted 2012-08-16; First posted 2012-08-21 (Estimated); Last update posted 2013-12-19 (Estimated); Status verified 2013-12

CONDITIONS: Fatigue
MeSH Terms: conditions — Fatigue

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Red Bull™ Sugar-Free Drink (Experimental): Red Bull™ Sugar-Free Drink: two (250mL) cans per day for 28 days
  Interventions: Other: Red Bull™ Sugar-Free Drink

INTERVENTIONS:
Other: Red Bull™ Sugar-Free Drink — Red Bull™ Sugar-Free Drink two (250mL) cans per day for 28 days

SUMMARY:
The purpose of this research study is to find out if Red Bull™ Sugar-Free Drink can reduce fatigue in prostate cancer patients receiving LHRH agonist therapy.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed prostate cancer
* Currently receiving LHRH-agonist therapy for greater than 6 months
* Measurable fatigue, defined as a score of ≥ 2 on the Bruera global fatigue severity scale
* Able to swallow Red Bull™ Sugar-Free Drink
* Life expectancy of at least 1 year
* Able to read and write in English
* Willing to limit consumption of alcohol to one drink per day

Exclusion Criteria:

* Current malignancy or received treatment for a previous malignancy within the last 3 years other than prostate cancer (exceptions are superficial bladder cancer or non-melanoma skin cancer)
* Myocardial infarction within past 6 months
* Any unstable serious co-existing medical condition(s) including but not limited to unstable or poorly controlled coronary artery disease, chronic atrial fibrillation, uncontrolled hypertension, uncontrolled diabetes, severe bleeding diseases or immune disorders
* Evidence of drug or alcohol abuse
* Known hypersensitivity to caffeine
* Known history of liver and kidney insufficiencies
* Known contraindications to Red Bull™ use

Ages: 18 Years to 85 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2012-07; Primary Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Reduction in overall fatigue as measured by Bruera global fatigue severity scale. | Within 4 days after completion of intervention (28 days of Red Bull™)

SECONDARY OUTCOMES:
Overall improvement in quality of life as measured by the Medical Outcomes Study Short-Form (SF-36) | Within 4 days after completion of intervention (28 days of Red Bull™)

CONTACTS AND LOCATIONS:
Overall Officials: Neil Fleshner, MD, FRCSC, MPH, Principal Investigator — University Health Network, Toronto
Locations (1):
- University Health Network, Toronto, Ontario, Canada